CLINICAL TRIAL: NCT01242722
Title: Evaluation of Left Ventricular Autothreshold, Phase Two
Acronym: ELEVATE 2
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ELEVATE 2.0
Record Dates: First submitted 2010-11-12; First posted 2010-11-17 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Heart Failure
Keywords: Heart failure; auto threshold; pacing; CRT-D recipients; Left Ventricular (LV) evoked response signals
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Two experimental and/or intervention groups under 1 arm.
  Interventions: Device: CRT-D

INTERVENTIONS:
Device: CRT-D — Cardiac pacing via a pulse generator and implanted intracardiac leads

SUMMARY:
This study will collect data, from an implanted Cardiac Resynchronization Therapy-Defibrillator (CRT-D) device, to further evaluate a new feature for future heart failure devices.

DETAILED DESCRIPTION:
ELEVATE 2.0 is an acute, prospective, multi-center, feasibility study randomized within patient test sequence and pulse width, designed to characterize the performance of the Left Ventricular Auto Threshold (LVAT) feature.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a COGNIS CRT-D device implanted for at least 24 hours, with or without a right atrial lead
* Patients who have an active LV bipolar lead
* Patients who have an active right ventricular (RV) defibrillation lead
* Patients who are willing and capable of participating in all testing associated with this Clinical Investigation
* Patients who are age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Patients who have a COGNIS CRT-D that has less than or equal to one year of battery life remaining
* Patients who are pacemaker-dependent
* Patients who will not tolerate a pacing pause of up to 6 seconds
* Patients who have a unipolar LV pace/sense lead, unless the patient has any commercially available epicardial leads with at least two electrodes (from one or more leads)
* Patients with pre-existing leads other than those specified in this investigational plan
* Patients with a pre-existing unipolar pacemaker
* Patients who are unable or unwilling to maintain a supine or sitting position for 40-50 minutes
* Patients enrolled in any concurrent study, without Boston Scientific written approval
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be a sample of patients with COGNIS CRT-D devices and bipolar LV leads.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Collect ventricular evoked response signals and CRT-D device data during LV only and Bi-ventricular (Bi-V) voltage step down pacing | At least 24 hours post CRT-D implant
  The primary objective of this study is to collect real-time signals during LV pacing voltage step-down from patients with implanted COGNIS CRT-D devices in a follow-up setting. This data will be used to assess the stability of the LV evoked response electrogram signal and will be used in an offline assessment of the LVAT algorithm. One or two data points will be collected per patient in the trial. Patients must be at least 24 hours post implant of their COGNIS CRT-D device

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Ellenbogen, M.D., Principal Investigator — Virginia Commonwealth University Health System
Locations (1):
- Regional Cardiovascular Medical Center, Stuebenville, Ohio, United States